CLINICAL TRIAL: NCT00004873
Title: Taxotere-Cisplatin-5FU (TCF) Versus Taxotere-Cisplatin (TC) Versus Epirubicin-Cisplatin-5FU (ECF) as Systemic Treatment for Advanced Gastric Carcinoma: A Randomized Phase II Trial
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: SAKK 42/99; SWS-SAKK-42/99; EU-99021
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Gastric Cancer
Keywords: stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin; Docetaxel; Epirubicin; Fluorouracil

INTERVENTIONS:
Drug: cisplatin
Drug: docetaxel
Drug: epirubicin hydrochloride
Drug: fluorouracil

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which combination chemotherapy regimen is most effective in treating advanced stomach cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of different regimens of combination chemotherapy in treating patients who have advanced stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy and tolerability of docetaxel, cisplatin, and fluorouracil (TCF) versus docetaxel and cisplatin (TC) versus epirubicin, cisplatin, and fluorouracil (ECF) in patients with advanced gastric carcinoma.
* Compare the time to treatment failure, time to progression, and survival in this patient population treated with these regimens.
* Compare the quality of life during the treatment period and after failure in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, performance status (0 vs 1), and liver involvement (yes vs no). Patients are randomized to one of three treatment arms.

* Arm I: Patients receive epirubicin IV bolus and cisplatin IV over 4 hours on day 1 plus fluorouracil IV continuously on days 1-21.
* Arm II: Patients receive docetaxel IV over 1 hour and cisplatin IV over 4 hours on day 1.
* Arm III: Patients receive docetaxel and cisplatin as in arm II and fluorouracil as in arm I.

Treatment regimen is repeated every 3 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed before randomization; at day 1 of courses 2, 4, and 6; and one month after treatment failure.

Patients with complete response or partial response are followed monthly for 3 months.

PROJECTED ACCRUAL: Approximately 111 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed gastric carcinoma not amenable to curative surgery or in relapse after primary surgical resection

  * Locally advanced disease (i.e., measurable locoregional lymph nodes) OR
  * Metastatic disease
* Bidimensionally measurable disease

  * At least 10 mm X 20 mm by chest x-ray or physical examination
  * At least 10 mm X 10 mm by CT scan
* No CNS metastasis

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Performance status:

* 0-1

Life expectancy:

* Greater than 12 weeks

Hematopoietic:

* WBC count at least 4,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 5 times ULN

Renal:

* BUN normal
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* No severe hypercalcemia

Cardiovascular:

* No unstable cardiac disease requiring treatment
* No congestive heart failure
* No angina pectoris even if medically controlled
* No significant arrhythmias
* No prior myocardial infarction unless ejection fraction at least 50% by MUGA scan or echocardiogram

Neurologic:

* No prior significant neurologic or psychiatric disorders, including psychotic disorders, dementia or seizures that would preclude study
* No peripheral neuropathy of any origin (alcohol, etc.) greater than grade 1

Other:

* Fertile patients must use adequate contraception
* No prior malignancy except basal cell skin cancer or adequately treated carcinoma in situ of the cervix
* No active uncontrolled infection
* No other serious illness or medical condition that would preclude study participation
* No contraindication to corticosteroid use

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior palliative chemotherapy
* At least 12 months since prior adjuvant or neoadjuvant chemotherapy
* No prior taxanes
* Prior fluorouracil allowed in bolus form only
* Prior cumulative dose of adjuvant or neoadjuvant cisplatin no greater than 300 mg/m2

Endocrine therapy:

* Prior or concurrent prednisone (or equivalent) allowed for prophylaxis, acute hypersensitivity reactions, or chronic therapy (greater than 6 months) at doses no greater than 20 mg

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* No other concurrent experimental drugs
* No other concurrent anticancer therapies
* At least 30 days since treatment in prior clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Roth, MD, Study Chair — Hopital Cantonal Universitaire de Geneve
Locations (1):
- Hopital Cantonal Universitaire de Geneva, Geneva, Switzerland

REFERENCES:
- [Result] Roth AD, Fazio N, Stupp R, Falk S, Bernhard J, Saletti P, Koberle D, Borner MM, Rufibach K, Maibach R, Wernli M, Leslie M, Glynne-Jones R, Widmer L, Seymour M, de Braud F; Swiss Group for Clinical Cancer Research. Docetaxel, cisplatin, and fluorouracil; docetaxel and cisplatin; and epirubicin, cisplatin, and fluorouracil as systemic treatment for advanced gastric carcinoma: a randomized phase II trial of the Swiss Group for Clinical Cancer Research. J Clin Oncol. 2007 Aug 1;25(22):3217-23. doi: 10.1200/JCO.2006.08.0135. PMID 17664469